CLINICAL TRIAL: NCT01881412
Title: Optimizing Discharge After Emergency Department Visits for Children With Uncontrolled Asthma
Brief Title: Inhaled Steroids at Discharge After Emergency Department Visits for Children With Uncontrolled Asthma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding complete
Sponsor: Rhode Island Hospital (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACP-231928-N; ACP-231928-N (Other Grant/Funding Number: American Lung Association)
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2018-04

CONDITIONS: Asthma
Keywords: Asthma; Children; Inhaled Corticosteroids; Emergency Department
MeSH Terms: conditions — Asthma; Emergencies | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled corticosteroid (fluticasone) (Experimental): Child receives: 1) standardized asthma discharge instructions, and the intervention which is 2) inhaled corticosteroid prescription with accompanying instructions.
  Interventions: Drug: fluticasone; Other: Standard Asthma Discharge Instructions
- Routine Asthma Care (Placebo Comparator): Child receives: 1) Standard Asthma Discharge Instructions. No intervention in this arm (placebo controlled)
  Interventions: Other: Standard Asthma Discharge Instructions

INTERVENTIONS:
Drug: fluticasone — During discharge, the study MD/nurse informs the family that the child has been randomized to the inhaled corticosteroid (ICS) group, and will be prescribed fluticasone to help control the asthma. The families preferred pharmacy is determined and a prescription for a fluticasone multi-dose inhaler (MDI) provided. Dosing follows the NHLBI asthma guidelines for low dose ICS in this age group (88 mcg administered twice per day, dispense one inhaler, 3 refills). In addition to standard asthma discharge instructions, the family receives specific instructions for ICS administration, possible side effects of medication use, and distinction between controller and quick-relief rescue medications. Parents are instructed to discuss with their primary care provider the length of ICS use.
  Other Names: inhaled corticosteroid
  Arms: Inhaled corticosteroid (fluticasone)
Other: Standard Asthma Discharge Instructions — Study MD or nurse provides asthma discharge instructions using a standardized checklist. The topics covered include 1) description of asthma manifestations related to current visit, 2) signs of respiratory distress family should be looking for, 3) instructions to follow up with the child's primary care provider within one week, 4) provision and review of an asthma action plan, 5) provision of a spacer device to be used with inhalers (if family does not already possess), and 6) smoking cessation advice. (if indicated)

SUMMARY:
Many children have asthma and this causes problems with their health. A lot of children with uncontrolled asthma use emergency departments for asthma care, and so this is an ideal place for an intervention for these children. One intervention is prescribing inhaled steroids to children with uncontrolled asthma, but currently this is rarely done in the emergency department. Inhaled steroids have been shown to be good at making children better long-term when they have uncontrolled asthma.

This study identifies children in the emergency department with uncontrolled asthma using a tool called the Pediatric Asthma Control and Communication Instrument (PACCI). If children meet criteria for uncontrolled asthma they will be randomly assigned to either: 1) routine asthma care which includes close follow up with their doctor or 2) prescribing of an inhaled corticosteroid from the emergency department. The investigators hypothesize that children who are prescribed inhaled steroids for uncontrolled asthma from the emergency department will have better 6 month asthma control than children who receive routine asthma care.

DETAILED DESCRIPTION:
Specific aim 1 - An ED-based RCT to determine if ICS prescription in children identified using the PACCI as having uncontrolled asthma results in less asthma morbidity compared to routine asthma care. We hypothesize that children receiving ICS prescriptions will have fewer unscheduled health care use for asthma exacerbations (doctor's office visits, ED visits, or hospitalizations), and greater quality of life.

Specific aim 2 - Thematic analysis of interviews with parents who are adherent versus non-adherent with ICS prescription filling and use to determine the factors associated with adherence. We hypothesize that factors will include: 1) Parent beliefs about the chronic versus episodic nature of asthma, 2) Parent's knowledge of benefits and risks of ICS, and 3) Provision and use of an asthma action plan.

ELIGIBILITY:
Inclusion Criteria:

* 3 - 12 years of age
* child has asthma diagnosed by a doctor based on parental/caregiver report
* child is not already properly using an ICS or being discharged with an ICS

Exclusion Criteria:

* The child has previously participated in this study
* The child has major co-morbid disease of the heart or lungs (examples include cystic fibrosis, heart disease, muscular dystrophy and cerebral palsy with immobility. It does not include allergic rhinitis or a history of respiratory infections such as pneumonia or bronchiolitis.
* The child's parents/caregivers do not speak English
* The child is not going to be discharged from the emergency department (e.g. hospitalization)

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aris C Garro, MD, MPH, Principal Investigator — Brown University and Rhode Island Hospital
Locations (1):
- Rhode Island Hospital / Hasbro Children's Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Availability on request
Supporting Information: Study Protocol, ICF
Time Frame: Data currently available on request
Access Criteria: Requests will be reviewed by the study investigators for appropriateness

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled Corticosteroid (ICS): Child receives: 1) asthma discharge instructions, and 2) ICS prescription.
  Asthma Discharge Instructions include 1) describing asthma symptoms, 2) signs of respiratory distress, 3) instructions to visit the primary care provider within a week, 4) provision/review of asthma action plan, 5) providing an aerochamber device (if necessary) and 6) smoking cessation advice if indicated.
  The family is also told that the child has been randomized to be prescribed an ICS to help control the asthma. Prescribing follows the NHLBI asthma guidelines for low dose ICS in this age group with 3 refills provided. In addition to standard asthma discharge instructions, the family receives specific instructions for ICS administration, possible side effects of ICS use, and teaching about controller and quick-relief rescue medications. Parents are instructed to discuss with their primary care provider the length of ICS use.
- Routine Asthma Care: Child receives: 1) Standard Asthma Discharge Instructions. No intervention in this arm (placebo controlled)
  Asthma Discharge Instructions include 1) describing asthma symptoms, 2) signs of respiratory distress, 3) instructions to visit the primary care provider within a week, 4) provision/review of asthma action plan, 5) providing an aerochamber device (if necessary) and 6) smoking cessation advice if indicated.
Period: Overall Study
Arm/Group | Inhaled Corticosteroid (ICS) | Routine Asthma Care
Started | 59 | 59
Completed | 49 | 57
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Corticosteroid (ICS) | Routine Asthma Care | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (2.4) | 6.4 (2.3) | 6.3 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 43 | 37 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 14 | 38
  Black | 7 | 13 | 20
  Hispanic | 20 | 19 | 39
  Mixed race / other | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: Quality-of-life Using the Integrated Therapeutics Group Child Asthma Short Form
Description: The Integrated Therapeutics Group Child Asthma Short Form (ITG-CASF) has been validated in the ED setting for children 2 to 17 years old, is reliable (Cronbach's α =0.70), and can be administered by telephone. Each item is rated on a 5-point scale. Each response is scaled as a percentage of the maximum response, and the total score is the maximum percentage based on the number of questions answered. The scores range from 0 (minimum) - 100 (maximum), with higher scores reflecting better quality of life. The change in ITG-CASF scores for children with improved overall clinical status are 10 points higher than when children have not improved.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Inhaled Corticosteroid (Fluticasone): Child receives: 1) standardized asthma discharge instructions, and the intervention which is 2) inhaled corticosteroid prescription with accompanying instructions.
  fluticasone: The families preferred pharmacy is determined and a prescription for a fluticasone multi-dose inhaler (MDI) provided. Dosing follows the NHLBI asthma guidelines for low dose ICS in this age group (88 mcg administered twice per day, dispense one inhaler, 3 refills).
  Standard Asthma Discharge Instructions: 1) description of asthma manifestations related to current visit, 2) signs of respiratory distress family should be looking for, 3) instructions to follow up with the child's primary care provider within one week, 4) provision and review of an asthma action plan, 5) provision of a spacer device to be used with inhalers (if family does not already possess), and 6) smoking cessation advice. (if indicated)
Arm/Group | Inhaled Corticosteroid (Fluticasone) | Routine Asthma Care
Number analyzed (Participants) | 59 | 59
score on a scale | 90 (14) | 84 (16)

2. Secondary Outcome: ED Visits for Asthma
Description: Emergency department visits for asthma over a 6 month period by parent report.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Inhaled Corticosteroid (Fluticasone) | Routine Asthma Care
Number analyzed (Participants) | 59 | 59
visits | .37 (1) | 0.56 (0.8)

3. Secondary Outcome: Primary Care Visits for Well Checks
Description: Primary care visits well checks over a 6 month period by parent report.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Inhaled Corticosteroid (Fluticasone) | Routine Asthma Care
Number analyzed (Participants) | 59 | 59
visits | 1 (1.1) | 0.6 (0.8)

4. Secondary Outcome: Hospitalizations for Asthma
Description: Hospitalizations for asthma over a 6 month period by parent report.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Inhaled Corticosteroid (Fluticasone) | Routine Asthma Care
Number analyzed (Participants) | 59 | 59
Hospitalizations | .06 (.32) | .05 (.23)

5. Secondary Outcome: Unscheduled Primary Care Visits
Description: Unscheduled primary care visits for asthma over a 6 month period by parent report.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Inhaled Corticosteroid (Fluticasone) | Routine Asthma Care
Number analyzed (Participants) | 59 | 59
visits | .8 (1) | 1.7 (2.8)

6. Secondary Outcome: Oral Steroid Courses
Description: Oral steroid courses over a 6 month period by parent report.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Courses
Arm/Group | Inhaled Corticosteroid (Fluticasone) | Routine Asthma Care
Number analyzed (Participants) | 59 | 59
Courses | .54 (.87) | 0.7 (1.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Inhaled Corticosteroid (Fluticasone) | Routine Asthma Care
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT01881412/Prot_SAP_000.pdf